CLINICAL TRIAL: NCT03014947
Title: A Phase I, Randomized, Double-Blind, Parallel-Group, Single-Dose Trial to Compare the Pharmacokinetics, Safety, Tolerability, and Immunogenicity of MSB11022, US-Reference Product, and EU-Reference Medicinal Product (Humira®) in Healthy Subjects
Brief Title: MSB11022 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fresenius Kabi SwissBioSim GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMR200588-001; 2014-000662-21 (EudraCT Number)
Record Dates: First submitted 2017-01-06; First posted 2017-01-09 (Estimated); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Healthy Subjects
Keywords: MSB11022; Humira®

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- MSB11022 (Experimental)
  Interventions: Drug: MSB11022
- US-licensed Humira (Active Comparator)
  Interventions: Drug: US-licensed Humira
- EU-approved Humira (Active Comparator)
  Interventions: Drug: EU-approved Humira

INTERVENTIONS:
Drug: MSB11022 — Subjects will receive single dose of 40 milligram (mg) MSB11022 as a subcutaneous injection in the lower abdomen on Day 1.
  Arms: MSB11022
Drug: US-licensed Humira — Subject will receive single dose of 40 mg US-licensed Humira as a subcutaneous injection in the lower abdomen on Day 1.
  Arms: US-licensed Humira
Drug: EU-approved Humira — Subject will receive single dose of 40 mg EU-approved Humira as a subcutaneous injection in the lower abdomen on Day 1.
  Arms: EU-approved Humira

SUMMARY:
This is a phase I, randomized, double-blind, parallel-group trial to compare Investigation Medicinal Product (IMP) MSB11022, US- Reference Product (RP), and EU- Reference Medicinal Product (RMP) (Humira®) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects and healthy female subjects of non-childbearing potential aged 18 to 55 years, inclusive.
* Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

* Concurrent or history infections such as opportunistic infections, including sepsis, pneumonia, and fungal infection.
* Individuals with history of tuberculosis or diagnosed with tuberculosis by interview, chest X-ray examination, or interferon-gamma release assay.
* Concurrent or history of demyelinating disease (multiple sclerosis, etc.).
* Concurrent or history of congestive cardiac failure.
* Concurrent or history of allergic symptoms such as asthma bronchial, drug-induced rash, and urticaria, which, in the judgment of the investigator, may affect participation in this clinical study.
* Concurrent or history of cardiac, hepatic, renal, gastrointestinal, respiratory, and/or hematological function disorders, which, in the judgment of the investigator or any of the sub investigators, may affect participation in this clinical study.
* Other protocol defined exclusion criteria could apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 237 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Primary: Area Under the Concentration-Time Curve From time Zero Extrapolated to Infinity (AUC [0-inf]) | Pre-dose 0 hour, post-dose 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 240, 336, 504, 672, 840, 1008, 1344, 1680 hours
Maximum Observed Serum Concentration (Cmax) | Pre-dose 0 hour, post-dose 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 240, 336, 504, 672, 840, 1008, 1344, 1680 hours
Area Under the Concentration-Time Curve From Time Zero to the Last Quantifiable Concentration (AUC [0-last]) | Pre-dose 0 hour, post-dose 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 240, 336, 504, 672, 840, 1008, 1344, 1680 hours

SECONDARY OUTCOMES:
Time to Reach Maximum Observed Serum Concentration (Tmax) | Pre-dose 0 hour, post-dose 4, 8 12, 24, 48, 72, 96, 120, 144, 168, 192, 240, 336, 504, 672, 840, 1008, 1344, 1680 hours
Apparent Volume of Distribution During the Terminal Phase (Vz/F) | Pre-dose 0 hour, post-dose 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 240, 336, 504, 672, 840, 1008, 1344, 1680 hours
Terminal Half-Life (t1/2) | Pre-dose 0 hour, post-dose 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 240, 336, 504, 672, 840, 1008, 1344, 1680 hours
Apparent Total Clearance (CL/F) | Pre-dose 0 hour, post-dose 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 240, 336, 504, 672, 840, 1008, 1344, 1680 hours
Number of Subjects With Injection Site Reactions | Baseline up to Day 71
Number of Subjects With Treatment-Emergent Adverse Events (AEs), Serious AEs (SAEs) and AEs Leading to Death | Baseline up to Day 71
Number of Subjects With Anti-drug Antibodies (ADA) for MSB11022 | Day 1 up to Day 71

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director

REFERENCES:
- [Result] Hyland E, Mant T, Vlachos P, Attkins N, Ullmann M, Roy S, Wagner V. Comparison of the pharmacokinetics, safety, and immunogenicity of MSB11022, a biosimilar of adalimumab, with Humira((R)) in healthy subjects. Br J Clin Pharmacol. 2016 Oct;82(4):983-93. doi: 10.1111/bcp.13039. Epub 2016 Jul 28. PMID 27285856
- [Derived] Huizinga TWJ, Torii Y, Muniz R. Adalimumab Biosimilars in the Treatment of Rheumatoid Arthritis: A Systematic Review of the Evidence for Biosimilarity. Rheumatol Ther. 2021 Mar;8(1):41-61. doi: 10.1007/s40744-020-00259-8. Epub 2020 Dec 1. PMID 33263165